CLINICAL TRIAL: NCT05509101
Title: Improving Myoelectric Prosthetic and Orthotic Limb Control Using Predictive Regression Algorithms and High-count Surface Electrodes
Brief Title: Improving Myoelectric Prosthetic and Orthotic Limb Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jacob George, Assistant Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB_00098851
Record Dates: First submitted 2022-08-15; First posted 2022-08-19 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Hemiparesis
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinically Available Control Algorithm (MyoPro) (Active Comparator): Binary control of the orthosis is based on a clinically available control algorithm. This condition serves as a control. Participants will use a commercially available device, the MyoPro.
  Interventions: Other: commercially available control algorithm
- High-Density EMG Control Algorithm (Experimental): Control of the orthosis is based on residual muscle activity mapped to intended movement using advanced predicted algorithms. This condition is a novel algorithm and serves as the experimental condition.
  Interventions: Other: experimental control algorithm

INTERVENTIONS:
Other: commercially available control algorithm — Control of the prosthesis/orthosis is based on clinical standard of care using commercially available control algorithms.
  Arms: Clinically Available Control Algorithm (MyoPro)
Other: experimental control algorithm — Control of the orthosis is based on residual muscle activity mapped to intended movement using high density electromyography and artificial intelligence control algorithms.
  Arms: High-Density EMG Control Algorithm

SUMMARY:
The purpose of this study is to improve control of myoelectrically-controlled advanced orthotic devices (an exoskeleton device that use the body's muscle signals to drive movements of a robotic brace) by using advanced predictive decode algorithms, and the use of high count (> 8) surface electromyographic (sEMG) electrodes.

DETAILED DESCRIPTION:
This study looks to improve control of myoelectrically-controlled advanced powered orthoses (orthoses that use the body's muscle signals to drive movements of a robotic exoskeleton) by using advanced predictive decode algorithms, and the use of high count (> 8) surface electromyographic (sEMG) electrodes.

ELIGIBILITY:
Inclusion Criteria:

* First-ever ischemic or hemorrhagic stroke
* Chronic Stroke (at least 6 months since onset)
* Chronic hemiparesis
* Functional range of motion for contralateral arm

Exclusion Criteria:

* Individuals who are currently Incarcerated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Box and Blocks Test (BBT) | while using the device (up to 2 hours)
  The Box and Blocks test is performed using the orthotic device under each condition. The individual puts on the device for a maximum of two hours. During that time wearing the device, they will use two different algorithms for controlling the device to complete the Box and Blocks Test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States